CLINICAL TRIAL: NCT00429624
Title: Randomized Controlled Trial of Chiropractic Manipulation Versus Medical Therapy for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Foundation for Chiropractic Education and Research (FCER) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 94-0085
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2007-01

CONDITIONS: Neck Pain
Keywords: Neck Pain; Chiropractic manipulation; Randomized controlled trial
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Chiropractic; Acetaminophen

INTERVENTIONS:
Procedure: Chiropractic manipulation
Drug: acetaminophen

SUMMARY:
The purpose of this study is to determine whether chiropractic manipulation or medical therapy is effective in the treatment of chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a common complaint, approximately 10% of the population have neck pain. Many modalities are used to treat neck pain, but no therapy has been found to be clearly superior. We conducted a randomized controlled study of chiropractic manipulation versus medical therapy for chronic neck pain.

Subjects (n=70) with neck pain for more than 3 months but with no evidence of radiculopathy or myelopathy were randomized. Both groups were instructed to do neck exercises and use heat daily. The chiropractic group received 12 standardized manipulations over 6 weeks. Nurses saw the medical group on the same visit schedule and received acetaminophen 1,000 milligrams four times a day as needed. Blinded observer performed all measurements. The primary outcome measure was the Neck Disability Index (NDI). Secondary measures were pain via a visual analogue scale, global via Medical Outcome Study Short Form and range of motion via Cybex electronic inclinometer.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain for more than 3 months

Exclusion Criteria:

* Cervical radiculopathy or myelopathy
* Contraindications to cervical manipulation: metastatic cancer, coagulation disorder, cervical spine abnormalities, neuromuscular disease
* Medical contraindications: uncontrolled hypertension, active coronary artery disease, history of cerebral vascular disease, alcohol or drug dependency, acetaminophen allergy
* Active litigation involving neck pain
* Medical or Chiropractic treatment within the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 1994-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index scale 0-30, clinically significant difference is a change greater than or equal to 5

CONTACTS AND LOCATIONS:
Overall Officials: David J Tanaka, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States